CLINICAL TRIAL: NCT02609360
Title: Effects of Different Crystalloid Solutions for Extra-corporeal Membrane Oxygenator (ECMO) Priming
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1897
Record Dates: First submitted 2015-11-07; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Acute Respiratory Failure
Keywords: Acute Respiratory Failure; ARDS; ECMO; Lung transplantation; Acid-Base Equilibrium
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.9% NaCl (Active Comparator): Circuit priming will be performed with 0.9% NaCl solution
  Interventions: Other: Priming of ECMO circuit with 0.9% NaCl
- Ringer Lactate (Active Comparator): Circuit priming will be performed with Ringer Lactated
  Interventions: Other: Priming of ECMO circuit with Ringer Lactate
- Balanced Solution (Experimental): Circuit priming will be performed with a Balanced Solution created by mixing 0.9% NaCl, Sodium bicarbonate (8.4%) and injectable sterile water, in order to obtain a solution with constant sodium concentration (140 mEq/l) and SID equal to patient's bicarbonate level.
  Interventions: Other: Priming of ECMO circuit with Balanced Solution

INTERVENTIONS:
Other: Priming of ECMO circuit with 0.9% NaCl — 0.9% NaCl as priming crystalloid solution
  Arms: 0.9% NaCl
Other: Priming of ECMO circuit with Ringer Lactate — Ringer Lactate as priming crystalloid solution
  Arms: Ringer Lactate
Other: Priming of ECMO circuit with Balanced Solution — Balanced Solution as priming crystalloid solution
  Arms: Balanced Solution

SUMMARY:
Crystalloid solutions modify acid-base equilibrium according to their electrolyte composition. Moreover, it has been suggested that these alterations are generated by the difference between the solution strong ion difference (SID) and the plasma bicarbonate level. An increased risk of acute kidney injury and renal replacement therapy has been associated to the infusion of chloride rich crystalloids. This study aims to compare, in patients with acute respiratory failure undergoing ECMO support, the effects on acid-base status and renal function of crystalloids commonly employed for circuit priming to a balanced solution created with a SID equal to patients' bicarbonate level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Respiratory Failure in need for ECMO treatment

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Variation in Acid-Base Equilibrium (Base Excess) | First 24 hours after ECMO start

SECONDARY OUTCOMES:
Variation in Acid-Base Equilibrium (pH) | First 24 hours after ECMO start
Variation in Renal Function | First 24 hours after ECMO start

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Caironi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy